CLINICAL TRIAL: NCT06943859
Title: Ketamine for the Treatment of Opioid Use Disorder
Brief Title: Ketamine for Opioid Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Peter Manza, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00114026
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder; ketamine; craving; treatment adherence; methadone
MeSH Terms: conditions — Opioid-Related Disorders; Treatment Adherence and Compliance | interventions — Therapeutics; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment with Ketamine (Experimental): Individuals will receive four doses spaced 1-6 days apart of 0.75mg/kg of intramuscular ketamine (n=25) over a period of two weeks.
  Interventions: Drug: Treatment with Ketamine
- Treatment with Very Low Dose Ketamine (Active Comparator): Individuals will receive four doses spaced 1-6 days apart of an intramuscular ketamine (0.1mg/kg) (n=25) over a period of two weeks.
  Interventions: Drug: Treatment with Very Low Dose Ketamine

INTERVENTIONS:
Drug: Treatment with Ketamine — Participants will receive four doses of ketamine spaced 1-6 days apart of 0.75 mg/kg intramuscular ketamine (n=25) for two weeks (first ketamine session must occur no later than 28 days post-intake). Individuals will be monitored for two hours post-dose by a clinician.
  Arms: Treatment with Ketamine
Drug: Treatment with Very Low Dose Ketamine — Participants will receive four doses of very low dose ketamine (0.1mg.kg) (n=25) spaced 1-6 days apart for two weeks (first ketamine session must occur no later than 28 days post-intake). Individuals will be monitored for two hours post-dose by a clinician.
  Arms: Treatment with Very Low Dose Ketamine

SUMMARY:
The goal of this clinical trial is to learn if ketamine works to reduce craving for opioids in adults entering methadone treatment for opioid use disorder. The main questions it aims to answer are:

* Does ketamine reduce craving for opioids in patients with opioid use disorder?
* Does ketamine reduce symptoms of opioid withdrawal such as depression, pain, and poor sleep quality?
* Do patients who take the low dose ketamine stay in methadone treatment longer, and/or have better treatment outcomes than those given the very low dose?

Researchers will compare two low doses of ketamine to see if ketamine works to reduce craving for opioids in adults entering methadone treatment for opioid use disorder.

Participants will:

* Be given a low dose or a very low dose of ketamine 4 times over a period of 2 weeks
* Visit the clinic weekly and monthly for checkups and tests for 90 days post-intake

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years old
2. Recent history (most recent 2 weeks prior to clinic intake) of routine use of illicit opioids, 5+ times/week
3. Fulfillment of DSM-5/ICD-10 criteria for moderate-to-severe opioid use disorder
4. Acceptance into methadone treatment for opioid use disorder within the past 21 days at the time of screening
5. Adherence to lifestyle requirements for participation

Exclusion Criteria:

1. Routine use of prescribed medications for OUD (5+ days/week) for longer than the 14 days leading up to clinic intake
2. Pregnant and/or breastfeeding
3. **Stage 2 Hypertension, defined by a systolic blood pressure (SBP) > 140mmHg or a diastolic blood pressure (DBP) > 90 mmHg
4. Abnormal oxygen saturation or abnormal heart rate (i.e. O2 saturation <95%, or HR <60 or >100bpm)
5. Clinically significant abnormal findings for which study participation is deemed unsafe
6. Severe mental illness or psychiatric disorder for which study participation is deemed unsafe (except for depression, PTSD, and substance use disorder)
7. **ALT/AST > 3 x Upper Limit of Normal (ULN), ALP 2 x ULN, or total bilirubin > 1.5 x ULN. Source: Labs
8. History of hypersensitivity to ketamine
9. Suicidal ideation with a plan or intent or suicidal behaviors as reflected in Columbia-Suicide Severity Rating Scale (C-SSRS)
10. Recent homicidal ideation or violent behaviors
11. Concomitant daily use of medications with significant CYP2B6 and CYP3A4 inhibition or induction effects that can interfere with metabolism of ketamine
12. Advanced cardiopulmonary disorders, including stroke, cardiac arrest, and myocardial infarction in the past year
13. History of aneurysmal vascular disease or dissection (including thoracic and abdominal aorta, intracranial, and peripheral arterial vessels) or arteriovenous malformation
14. **Clinically significant EKG abnormalities.
15. Current significant use (>3 days/week) of barbiturates, sedative hypnotics, benzodiazepines, ketamine, or PCP (prescribed or illicit)

    * NOTE: Due to time constraints in the study design, these exclusion criteria do not need to be met before the initial consent to participate. This criterion only needs to be established prior to the first ketamine session. Individuals that are initially enrolled and subsequently do not qualify due to severe hepatic impairment will be considered screen failures and withdrawn from the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Tonic craving (FORCAST) total scores | Collected at baseline, weekly, 30-, 60-, and 90 days post-intake
  Faceted Opioid Research Craving Assessment for Substance use Treatment (FORCAST): A 26-item assessment of tonic craving that the person reports having felt over the prior one or two weeks. Participants indicate how much they disagree or agree with each statement on a scale that ranges from 0-6, with 0 representing "strongly disagree", 3 representing "neither agree nor disagree", and 6 representing "strongly agree". Higher scores indicate higher levels of craving. The minimum score is 0, and the maximum scores for each of the subscales are as follows:
  Preoccupation: 24 Negative Reinforcement: 30 Positive Reinforcement: 24 Motivation: 30 Lack of control: 24 Uneasiness: 24
  Maximum total score for all subscales = 156

SECONDARY OUTCOMES:
Severity of depression symptoms | Completed at baseline, weekly, 30-, 60-, and 90 days post-intake
  Montgomery-Asberg Depression Rating Scale (MADRS): a 10-item questionnaire of depression severity. The total score ranges from 0-60, with scores of 0-6 considered normal (non-depressed), 7-19 indicative of mild depression, 20-34 indicative of moderate depression, and 35-60 indicative of severe depression. Item 10 on the instrument will be used to monitor any changes in suicidal ideation throughout the trial.
Cue-induced craving scores | Collected at Baseline, weekly following intake, 30-, 60-, and 90 days post-intake
  Cue Reactivity Paradigm: our drug cue reactivity paradigm will be designed to elicit an acute craving state. We will present a series of opioid cue images continuously (total time <5 min) via computer or tablet. Cues will be personalized based on each individual's drug use history as derived from baseline clinical assessments. For example, if a participant had no history of intravenous drug injection, we will not present opioid cue images containing injection paraphernalia like needles and instead will present images with opioid pills and/or powder. At the end of each one-minute session, participants will be asked to rate, on a scale of 1-10, "How much did you like the images you saw?", "How much do you want to use right now?", "How much do you want to avoid using right now?", "How much control do you feel you have over using right now" and "What is the maximum amount you would pay right now for a single dose of what you saw?"
Chronic pain ratings | Collected at Baseline, weekly following intake, 30-, 60-, and 90 days post-intake
  Pain Brief Scale (PEG): A 3-item measure of past-week average pain intensity (P), interference with enjoyment of life (E), and interference with general activity (G).
Number of methadone doses received at 90 days post-intake | Collected through 90 days post-intake
  Study team will have access to clinic records to assess the number of methadone doses patients have received at 90 days post-intake
Sleep quality ratings | PSQI collected at Baseline and 30-, 60-, and 90 days post-intake
  Pittsburgh Sleep Quality Index (PSQI): A 19-item questionnaire assessing past-month sleep quality and disturbances. Seven component scores are generated: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for the 7 components yields one global score
Insomnia Symptoms | ISI collected at Baseline, weekly following intake, 30-, 60-, and 90 days post-intake
  Insomnia Severity Index (ISI): A five-item measure of current (past two weeks, or since last study visit) insomnia symptoms.
Sleep quality ratings on a Visual Analogue Scale (VAS) | SQS collected via daily optional EMAs through 90 days post-intake
  Modified Single Item Sleep Quality Scale (SQS): A self-administered questionnaire that incorporates a VAS delivered electronically. SQS directs the patient to rate the overall quality of sleep over a 7-day period (modified for our study to rate the overall quality of sleep the past night) on a scale of 1-10 considering how many hours of sleep they had, how easily they fell asleep, how often they woke up during the night (excluding bathroom trips), how often they woke up earlier than intended
Scores on a holistic measure of recovery | Collected at baseline and at 30-, 60-, and 90 days post-intake
  Substance Use Recovery Evaluator (SURE): A 21-item patient reported outcome measure of recovery from substance use disorder that has good face and content validity, acceptability and usability for people in recovery and is psychometrically valid.
Frequency of negative urine drug screens through 90 days post-intake | collected through 90 days post-intake
  Study team will have access to clinic drug screenings through 90 days post-intake

OTHER OUTCOMES:
Decision making test performance (risk and ambiguity tolerance) | collected weekly through 90 days post-intake via optional EMAs
  Choice under risk and ambiguity (CRA) decision making task: On each trial, participants choose between a guaranteed $1 and a lottery. Each lottery has 2 possible outcomes: v or $0, where v ranges from $1.20 to $13.20. On half of the trials, v could be received with 1 of 3 known probabilities (p: 25%, 50%, or 75%); on the other half, the probability information is occluded and thus incompletely known (the ambiguity context). There are 3 levels of ambiguity: low (24% unknown), medium (50% unknown), and high (74% unknown). In reality, the true underlying probability in ambiguity trials is fixed at 50%. Different combinations of v, risk level, and ambiguity level are presented for 30 trials total.
  A modified utility model will be used which can extract the following parameters from participant decisions on these trials:
  * risk tolerance
  * ambiguity tolerance
  * choice stochasticity
Methadone dose (mg) at 90 days post-intake | collected through 90 days post-intake
  Study team will have access to clinic records of methadone dose (mg) received by participant at 90 days post-intake
OUD treatment outcomes at 6-, 9-, and 12 months post intake | collected through 6-, 9-, and 12 months post intake
  Study team will have access to clinic records of methadone dose, number of methadone doses received, and frequency of negative drug screens though 12 months post intake

CONTACTS AND LOCATIONS:
Overall Officials: Peter Manza, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Addiction Programs and Affiliated Clinics, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided